CLINICAL TRIAL: NCT00150514
Title: A Placebo Controlled, Double-Blind, Randomised Study to Assess Efficacy of Sublingual Immunotherapy in Patients With Grass Pollen Allergy Through Assessment of Its Immunological Effects on the Mucosal Tissue of the Nose.
Brief Title: Effects of Sublingual Immunotherapy on Grasspollen Allergy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AB0103
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2005-09-08 (Estimated); Status verified 2003-11

CONDITIONS: Hayfever
Keywords: nasal biopsy grasspollen sublingual immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Nasal Lavage Fluid

INTERVENTIONS:
Drug: Oralgen
Procedure: Nasal biopsy
Procedure: Nasal washing
Procedure: Peak nasal inspiratory flow

SUMMARY:
The objective of the study is to document the objective immunological effects of SLIT on the nasal mucosa. Better understanding of these immunological pathways, in which this widely practised clinical therapy is likely to work, can only benefit the overall outcome of this, more patient friendly, therapy and it will demonstrate the effects of SLIT on the allergic reaction, with objective parameters, in the nasal tissues showing it to be a true etiological treatment of allergy.

DETAILED DESCRIPTION:
Double blind placebo controlled evaluation of the immunological effects (decrease of IgE specific cells and the decrease of Th2 mediator release, respectively increase of Th1 mediator release) of SLIT on the nasal mucosal tissue of adult humans with severe rhinocunjunctivitis due to grass pollen allergy.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older.
2. Patients known in general practice with documented clinical history of grass pollen allergy with moderate disease intensity as retrospectively derived from the use of symptomatic allergy medication during the previous grass pollen season, i.e. regular use of cromoglycates as nasal spray and/or eye drops, and/or regular use of anti histamine tablets or sprays and/or limited use of local acting or systemically administered corticosteroids.
3. Positive (ARTU) grass pollen specific skin prick test (despite negative RAST).

Exclusion Criteria:

1. Clinical history of severe asthmatic symptoms requiring inhalant therapy with daily pulmonary steroids during at least 3 months a year.
2. Symptomatic perennial allergic rhinitis. Meaning perennial allergy is allowed if the allergen is not present in patients' daily life (especially one month prior to provocation) and if they have no apparent symptoms of this perennial allergy.
3. Other seasonal allergic rhinitis are not allowed unless it is asymptomatic during the period of provocation.
4. The intention to subject the patient to surgery of the nasal cavity in the course of the study.
5. Previous immunotherapy.
6. Negative (ARTU) grass pollen specific skin prick test (despite positive RAST).
7. Contraindications to sublingual immunotherapy, i.e.:

   * Malignancies and serious disorders of the oral cavity
   * History of status asthmaticus and anaphylactic shock
   * Aggressively developing asthmatic symptoms
   * Serious chronic inflammations, chronic disorders associated with fever, particularly of the bronchial tubes
   * Irreversible, secondary changes in reactive organs (emphysema, bronchiectasis)
   * Auto immune diseases and immunodeficiency
   * Concurrent therapy involving immunosuppressives
   * Systemic and collagen diseases
   * Tuberculosis of the lung and tuberculosis
   * Serious psychological disorders
   * Documented hypersensitivity to glycerol
   * Pregnancy
   * Serious cardiovascular disease
   * Usage of b -blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38
Dates: Start 2002-01; Study Completion 2006-12

PRIMARY OUTCOMES:
Double blind placebo controlled evaluation of the immunological effects of SLIT on the nasal mucosal tissue of adult humans with sever

SECONDARY OUTCOMES:
I. Correlating immunological effects to a retrospective subjective complaint reduction.
II. Rescue medication decrease through SLIT.
III. Determining the effects of SLIT on decongestion.
IV. Assessment of treatment compliance.

CONTACTS AND LOCATIONS:
Overall Officials: K Ingels, MD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboud university hospital, Nijmegen, Gelderland, Netherlands